CLINICAL TRIAL: NCT03041909
Title: An Open Label Single Arm Extension Study to Further Evaluate the Safety, Tolerability and Treatment Response of GBT440 in Patients With Sickle Cell Disease Who Participated in the Phase 1 Study GBT440-001
Brief Title: An Extension Study to Further Evaluate the Safety, Tolerability of GBT440 in Patients With Sickle Cell Disease Who Participated in the Study GBT440-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GBT440-024
Record Dates: First submitted 2017-01-19; First posted 2017-02-03 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Single Arm / open label
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — Oral drug

SUMMARY:
This is an open label, single arm study which enrolled 5 subjects with SCD who previously participated in the GBT440-001 study (NCT02285088).

DETAILED DESCRIPTION:
This is an open label, single arm study which enrolled 5 subjects with SCD who previously participated in the GBT440-001 study (NCT02285088).

Dosing of study drug was 2 to 6 months, depending on subject's dose assignment in the last administration of study drug in GBT440-001 (NCT02285088).

The primary objective of the study was to evaluate the safety and tolerability of up to a total of 6 months dosing of subjects with SCD who participated in the GBT440-001 study (NCT02285088).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with SCD aged 18 to 60 years inclusive and >50 kg who have participated in the GBT440-001 study.
2. Subjects, who if female and of child bearing potential, agree to continue to use highly effective methods of contraception prior to enrollment in this study and for 3 months after the last dose of study drug.
3. Subjects, who if male are willing to continue to use barrier methods of contraception, prior to enrollment in this study to 3 months after the last dose of study drug.

Exclusion Criteria:

1. Subjects requiring chronic transfusion therapy.
2. Subjects receiving a blood transfusion within 30 days of enrollment in this study.
3. Female subjects who are pregnant, trying to become pregnant or lactating.
4. Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, or additional risk factors for torsades de pointe (e.g., heart failure, hypokalemia, personal or family history of long QTc interval).
5. Subjects who have a significant infection or known inflammatory process on admission to this study.
6. Subjects who have acute gastrointestinal symptoms at the time of admission (e.g. nausea, vomiting, diarrhoea, heartburn).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Lehrer-Graiwer, MD, Study Director — Global Blood Therapeutics, Inc.; Timothy Mant, FRCP, FFPM, Principal Investigator — Quintiles, Inc.
Locations (1):
- The BRC Research Facility, Floor 15 The Tower Wing, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Howard J, Hemmaway CJ, Telfer P, Layton DM, Porter J, Awogbade M, Mant T, Gretler DD, Dufu K, Hutchaleelaha A, Patel M, Siu V, Dixon S, Landsman N, Tonda M, Lehrer-Graiwer J. A phase 1/2 ascending dose study and open-label extension study of voxelotor in patients with sickle cell disease. Blood. 2019 Apr 25;133(17):1865-1875. doi: 10.1182/blood-2018-08-868893. Epub 2019 Jan 17. PMID 30655275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled in this study participated in GBT440-001 study (NCT02285088).
Pre-assignment Details: There was no screening period as subjects transitioned directly from the GBT440-001 study (NCT02285088).into this study.
Groups:
- GBT440 - 2 Months: These subjects received GBT440 for 2 months as these subjects received GBT440 for 4 months in GBT440-001 study (n=3) (NCT02285088).
- GBT440 - 6 Months: The subject received GBT440 for 6 months as this subject received placebo in GBT440-001 study (n=1) (NCT02285088).
- GBT440 - 4 Months: This subject received GBT440 for 4 months as the subject received GBT440 for 2 months in GBT440-001 study (n=1) (NCT02285088).
Period: Overall Study
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months
Started | 3 | 1 | 1
Completed | 3 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GBT440 - 2 Months: These subjects received GBT440 for 2 months as these subjects received GBT440 for 4 months in GBT440-001 study (NCT02285088) (n=3).
- GBT440 - 6 Months: The subject received GBT440 for 6 months as this subject received placebo in GBT440-001 study (NCT02285088) (n=1).
- GBT440 - 4 Months: This subject received GBT440 for 4 months as the subject received GBT440 for 2 months in GBT440-001 study (NCT02285088) (n=1).
- Total: Total of all reporting groups
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months | Total
Number analyzed (Participants) | 3 | 1 | 1 | 5
Age, Continuous [Mean (Full Range); unit: Years] | 35 [25 to 42] | 26 | 21 | 30 [21 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 3 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events During Dosing of GBT440 for up to 6 Months.
Description: The safety evaluation will include physical examinations, blood pressure, clinical laboratory tests (hematology, serum biochemistry) and adverse events.
Time Frame: 2 - 6 months
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months
Number analyzed (Participants) | 3 | 1 | 1
Participants | 2 | 1 | 1

2. Secondary Outcome: To Assess the Efficacy of GBT440 as Measured by Improvements in Anemia
Description: Data presented are hemoglobin value collected at specific time points.
Time Frame: 2 - 6 months
Measure: Number; unit: g/dL
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months
Number analyzed (Participants) | 3 | 1 | 1
g/dL | NA — Data is not reported due to participant privacy. | NA — Data is not reported due to participant privacy. | NA — Data is not reported due to participant privacy.

3. Secondary Outcome: To Observed Pharmacokinetics in Plasma and Whole Blood.
Description: Measure maximum plasma concentration (Cmax)
Time Frame: 2 - 6 months
Measure: Number; unit: ug/mL
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months
Number analyzed (Participants) | 3 | 1 | 1
ug/mL | NA — Data is not reported due to participant privacy. | NA — Data is not reported due to participant privacy. | NA — Data is not reported due to participant privacy.

4. Secondary Outcome: To Characterize the Effect of GBT440 on Hemolysis.
Description: Data presented for unconjugated bilirubin at specific time point.
Time Frame: 2 - 6 months
Measure: Number; unit: umol/L
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months
Number analyzed (Participants) | 3 | 1 | 1
umol/L | NA — Data is not reported due to participant privacy. | NA — Data is not reported due to participant privacy. | NA — Data is not reported due to participant privacy.

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | GBT440 - 2 Months | GBT440 - 6 Months | GBT440 - 4 Months
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBT440 - 2 Months (N=3) | GBT440 - 6 Months (N=1) | GBT440 - 4 Months (N=1)
Sickle Cell Anemia with Crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBT440 - 2 Months (N=3) | GBT440 - 6 Months (N=1) | GBT440 - 4 Months (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival Swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor and the PI will have to agree on any publications regarding the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03041909/Prot_SAP_000.pdf